CLINICAL TRIAL: NCT02802189
Title: The Effect of Integrated Neuromuscular Inhibition Technique in Combination With Therapeutic Exercise on Patients With Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, LYTRAS DIMITRIOS, PhD Candidate, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AristotleU
Record Dates: First submitted 2016-06-07; First posted 2016-06-16 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Neck Pain
Keywords: Chronic Mechanical Neck Pain; exercise; Integrated Neuromuscular Inhibition Technique
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise and INIT group (Experimental): The first group (experimental) followed the exersice programme in combination with the integrated neuromuscular inhibition technique (INIT).
  Interventions: Other: Exercise programme; Other: Integrated Neuromuscular Inhibition Technique application.
- exercise group (Active Comparator): The protocol for this group was identical to the previous group with the sole difference that the application of INIT was not included.
  At the end of the exercise programme, relaxing breathing exercise and gentle stretching was applied for 15 min
  Interventions: Other: Exercise programme

INTERVENTIONS:
Other: Exercise programme — Endurance and Resistant training exercise program (Duration: 45 minutes)
  * Muscle retraining of longus colli and endurance training of the deep cervical flexors.
  * Resistant exercises for the muscles involved in neck flexion, extension, side bending and rotation of the neck region. Isometric contractions exercises (20-70% of MVC) and resistant exercises (12-15RM).
  * Active ROM exercises for the neck muscles
  * Upper limbs exercises with resistant bands
  * Stretching exercises for the neck and upper limbs muscles
Other: Integrated Neuromuscular Inhibition Technique application. — Integrated Neuromuscular Inhibition Technique application.
  (Duration: 15min)
  The protocol was applied to the following muscles:
  * Upper border of the trapezius muscle
  * sternocleidomastoid
  * levator scapulae muscle
  * splenius capitis muscle
  Integrated Neuromuscular Inhibition Technique includes the combination of the following technique:
  * Ischemic compression
  * Muscle energy technique
  * Strain-counterstrain technique
  Arms: exercise and INIT group

SUMMARY:
The purpose of this study is to examine the combine effect of the integrated neuromuscular inhibition technique (soft tissue mobilization techniques protocol), in combination with the therapeutic exercise in patients with chronic mechanical neck pain in the sub-acute stage of symptoms, and to determine whether this combination substantially helps the faster and more efficient installation of adaptations of exercising.

DETAILED DESCRIPTION:
Neck pain is one of the most common and costly musculoskeletal disorders in Western societies, which witnesses high prevalence of repeatability and chronicity. In chronic mechanical neck pain, there are changes in the neck area, due to muscular imbalance between deep neck flexors (longus capitis and longus colli) and superficial flexors of the neck (sternocleidomastoid and anterior scalene). Therapeutic exercise plays a key role in the restoration of this muscle imbalance, comprising a combination of resistant and endurance training. The integrated neuromuscular inhibition technique (INIT) is a manual deactivation trigger points technique and includes the application of ischemic pressure and stretch, the muscle energy technique and the Strain-counterstrain technique.

The aim of the research is to investigate whether the application of INIT combined with exercise can reduce the time required to establish the benefits of training and improve faster and to a greater extent the clinical figure and the quality of life of patients with chronic neck pain.

Method. Single blind clinical trial lasting for 10 weeks, 40 participants (men/women) with chronic mechanical neck pain. Participants will be divided into two groups, following the same exercise program. The first group (experimental) will follow the exercise programme in combination with the integrated neuromuscular inhibition technique (INIT), while the second (active comparator) will apply the same program excluding the INIT technique. The subjective perception of pain by the visual analogue scale, the functionality related to neck pain with neck disability index, ppt of the neck muscles with pressure algometry, active range of motion with a bubble inclinometer, maximum isometric strength of neck muscles with a hand dynamometer, muscular fatigue of the flexors of the neck with special tests and the quality of life with the sf-36 questionnaire will be evaluated before, during and after the intervention, while follow-ups will take place one, three and six months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic neck pain with a duration of symptoms for at least three months
* Existence of at least one active or latent trigger point in any of the muscles: levator scapulae, upper trapezoid, and splenius capitis
* Patients whose neck pain has emerged as a result of a specific pathology, confirmed by radio-diagnostic tests (X-ray or MRI)
* Patients with a medical referral for physical therapy with the etiology of neck pain

Exclusion Criteria:

* Patients who are in the acute stage of symptoms
* Patients who have participated in any kind of treatment during the last three months (physiotherapy, massage, local injections of anesthetic blocks, etc.)
* Patients who have participated in an exercise program concerning their neck during the last six months
* Background of neck trauma and / or surgery in the neck region
* Inflammatory muscle diseases and joint infections, malignancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in subjective perception of neck pain with the visual analogue scale (VAS) | pre-treatment, Week: 2, 4, 6,10,14, 22, 34
  Pain intensity was assessed by the Visual Analog Pain Scale, which is a card with an uncalibrated scale ranging from zero to ten on the one side (with zero representing no pain and ten representing the worst pain in life) with each centimeter representing one pain level. The patient subjectively estimated his or her pain level by marking a vertical line on the uncalibrated scale between zero and ten. Then the exact value of pain intensity could be obtained with a single ruler. VAS is widely used as it is easy to implement and is characterized by good psychometric properties.
Changes in Pressure Pain threshold with pressure algometry | pre-treatment, Week: 2, 4, 6, 10, 14, 22, 34
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure that produces pain. PPT was assessed by a Wagner algometer. For the procedure of PPT measurement, the protocol recommended by Fischer was applied (Fisher, 1998). Pressure pain threshold was assessed over the upper border of the trapezius muscle halfway between the midline and the lateral border of the acromion, the levator scapulae muscle 2 cm above the lower insertion located in the upper medial border of the scapulae, Sternocleidomastoid muscle and to splenius capitis 2 cm lateral to the spinous processus of the axis.
Changes in functional capacity with Neck disability index questionnaire | pre-treatment, Week 6, 10, 14, 22, 34
  It is a self-reported ten-item scale. Each item assesses different neck pain complaints. Most of the items are related to restrictions in activities of daily living, and each item is expressed by 6 different assertions in the range 0-5, with 0 indicating no disability and 5 indicating the highest disability. The total score ranges from 0 to 50. Disability Index (NDI) has sufficient support in the literature, being the most commonly used to report neck pain. The Greek version of the questionnaire was used for this study.
Changes in maximum isometric strength of neck muscles with Manual Muscular Testing | pre-treatment, Week: 2, 4, 6,10,14, 22, 34
  Cervical flexion, extension, and side bending isometric strength were assessed using a calibrated Manual Muscular Testing device with the participants in supine and prone position.
Changes in Cervical Range of Motion with a bubble inclinometer | pre-treatment, Week: 2, 4, 6,10,14, 22, 34
  Cervical active range of motion was measured with a bubble inclinometer. Active cervical flexion, extension, and side bending range of motion were assessed gravity with Participants sitting in upright position.
Changes in deep flexors muscle endurance with craniocervical flexion test | pre-treatment, Week: 2, 4, 6,10,14, 22, 34
  The craniocervical flexion test (CCFT) is a clinical test of the anatomical action of the deep cervical flexor muscles, (longus capitis, and longus colli). It could be described as a test of neuromotor control. It includes the performance of five progressive stages of increasing craniocervical flexion range of motion. It is a low-load test performed in the supine position with the patient guided to each stage by feedback from a pressure sensor placed behind the neck (Chattanooga Stabilizer Pressure Biofeedback). While the test in the clinical setting provides only an indirect measure of performance, the construct validity of the CCFT has been verified in a laboratory setting by direct measurement of deep and superficial flexor muscle activity.
Changes in isometric endurance capacity of sternocleidomastoid and anterior scalene, with a handheld stopwatch | pre-treatment, Week: 2, 4, 6,10,14, 22, 34
  The isometric endurance of the sternocleidomastoid and anterior scalene was assessed through 2 isometric contractions, one with no additional resistance and the other one with a kind of resistance corresponding to 30% of the maximum isometric strength. Participants were in supine position. A biofeedback device, provided the subject with motivation (auditory stimulus) encourage them to keep the contraction as long as possible. A 2-inch velcro band was secured around the forehead. The appropriate weight was suspended from the headband, and participants were asked to support the weight while maintaining a neutral head position for as long as possible. The endurance test was terminated when the position of the head changed (contact with table). Endurance time was measured using a handheld stopwatch.

SECONDARY OUTCOMES:
Changes in quality of life with the sort form of SF-36 Health Survey | pre-treatment, Week: 10, 14, 22, 34
  For the evaluation of the intervention in the quality of life of the participants the short form of SF-36 Health Survey questionnaire was used. SF-36 consists of 36 questions, selected from the Medical Outcomes Study (MOS), which relate to eight different parameters of mental and physical health.

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, New Facilities, Thermi, Thessaloniki, Greece